CLINICAL TRIAL: NCT00268008
Title: Retrospective Review of Children and Adolescents Receiving Mechanical and Prosthetic Valves in the Aortic and Mitral Position 1976-2002
Brief Title: Children and Adolescents Receiving Mechanical and Prosthetic Valves
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-033
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: aortic valve replacement; mitral valve replacement; valvular stenosis; Ross procedure; Homograft valves; Bio-prosthetic valves; Mechanical valves
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The primary objective of this retrospective study of valve replacement is to document long-term survival and occurrence of valve related complications such as described in the literature; anticoagulant related bleeding event , thromboembolic events, subacute bacterial endocarditis (SBE), structural failure or deterioration , valve thrombosis, explantation and reimplantation with reason, death and death cause, and cerebrovascular accidents either permanent or transient in nature.

Secondary to this is the presumption that mechanical valves have a superior "life expectancy " to bio-prosthetic valves. We plan to look at the time of freedom from re-implantation from different types of valves, factoring in patient age, size ,defect and risk factors.

The information learned from this study may benefit future patients who undergo the Ross procedure by increasing our knowledge of safer and/or more effective techniques.

DETAILED DESCRIPTION:
Both Aortic and Mitral valves utilizing bio-prosthetic and/or mechanical valves have been placed in adults since the 1960s.The replacement of these valves in children and adolescents began some 10 years after the first adult valve replacement. The majority of valves replaced in the pediatric cohort are due to either stenosis (narrowing) or incompetancy of the native valve. Valvular stenosis in the pediatric patient is normally of congenital etiology, however, a small percentage can be acquired from an infectious process. Stenosis of a valve impedes blood flow through the native valve orifice. Ventricular enlargement, hemodynamic instability and /or other major organ congestion can ensue if left untreated. Dependant upon the severity of the stenosis and the onset of the dysfunction, intervention may be required at any age (newborn to adult). In order for patients to have adequate blood flow to the systemic circulation (the body), the diseased valve must be replaced. Children with native valve stenosis experience failure to thrive, frequent pneumonia, difficulty breathing and generally poor physical development.

If the stenosis is of a critical nature greatly affecting hemodynamics, infants require intervention in the first few days of life. In these patients, initially many of the stenotic valves can be opened in the heart catheterization lab with a procedure called a valvuloplasty. While this procedure does open the valve leaflet apparatus, close approximation of the leaflets is not achieved and a residual insufficiency or regurgitation is present. Most infant hearts can handle minimal resurgent volumes from the resulting cardiac chamber enlargement. It will be necessary to surgically replace the incompetent valve with a prosthetic valve as the child grows. If valvuloplasty is unsuccessful, surgical intervention is required to relive the valvular Stenosis and improve hemodynamics.

Heart valve insufficiency creates a resurgence of blood back into either the left atrium or ventricle causing increased cardiac workload and dilation of the respective chamber of the heart. Incompetence of the Aortic valve will eventually cause congestive heart failure and/or sudden death from arrhythmias.

The initial surgery is dependant on the size of the ventricle and any other concomitant defects the child may have. A ventricle that is too small to support circulation will not be changed by placement of a valve. These patients require staged surgeries for single ventricle palliative repairs. Two examples of congenital cardiac defects include aortic stenosis and cleft mitral valve. If the aortic valve is stenosed and both ventricles are of adequate size, a Ross procedure can be done, The Ross procedure uses the patient's resected native pulmonary valve and main pulmonary artery in place of the aortic valve and outflow tract. A cryo-preserved homograft is then placed in the native pulmonary artery position. This homograft can be implanted with or without a valve dependant upon the patient's size and/or native valve orifice. Mitral valve anomalies occur frequently in patients with Atrioventricular septal defects. With this congenital defect the mitral valve may be dysplastic, or has a cleft in the anterior valve leaflet. This affects the competency of the valve, allowing regurgitation of blood flow into the left atrium. This increased blood volume in the left atrium will eventually lead to pulmonary hypertension. Because of this risk , repair of Atrioventricular septal defect is normally done between the ages of six and twelve months. Repair of the mitral valve is done at that time, with the knowledge that mitral valve replacement will be likely in the child's future. Repair of a heart valve in a patient of any age is always preferable to replacement; in children this is especially true.

Availability of replacement valves in infant sizes are limited to bio-prosthetic or homograft. Cryo-preserved homografts are made from either porcine and cadaver valves. These are generally used for pediatric patients under the age of two years. Historically homografts develop a significant amount of stenosis/calcification at the suture site. In addition, as the child grows the homograft size remains fixed. Both problems require further replacement.

Implantation of mechanical valves in the older children and young adults is considered as a treatment alternative. However, mechanical valves have inherent complications secondary to the requirement of long-term anticoagulant therapy (blood thinners) and the risk of thromboembolic events. Structural malfunctions of the valve and growth of the patient result in the need for replacement of mechanical valves. Additionally, patient compliance and dosing management can be difficult to control.

ELIGIBILITY:
Inclusion Criteria:

* Valve replacement in the mitral or aortic position
* replacement at Children's Healthcare of Atlanta
* replacement between 1976 and 2002
* implants may be mechanical, bio-prosthetic or homograft

Exclusion Criteria:

* those who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300
Dates: Start 1976-01

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R. Kanter, MD, Principal Investigator — Emory Univ. SOM Cardiothoracic Surgery of Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States